CLINICAL TRIAL: NCT04986852
Title: A Phase II, Open-Label, Multicenter Study of Olinvacimab in Combination With Pembrolizumab in Patients With Metastatic Triple-Negative Breast Cancer
Brief Title: Olinvacimab With Pembrolizumab in Patients With mTNBC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Subject recruitment issues and follow-up study plans
Sponsor: PharmAbcine (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMC_TTAC-0001_06 / KEYNOTE-C14; MK-3475-B37 (Other: Merck Sharp & Dohme Corp)
Record Dates: First submitted 2021-07-07; First posted 2021-08-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Triple-Negative Breast Cancer
Keywords: Olinvacimab; Pembrolizumab
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — olinvacimab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Patient will be assigned as sequentially with serial screening/ enrollment number.
Masking Description: It is open label study, so investigator and participant can know what is treated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olinvacimab (TTAC-0001) 16 mg/kg and Pembrolizumab (Keytruda®) 200 mg (Experimental): * Olinvacimab (TTAC-0001) 16 mg/kg on D1, D8 and D15
  * Pembrolizumab (Keytruda®) 200 mg on D1 Cycle: 3 weeks (21 days per cycle)
  Interventions: Drug: Olinvacimab

INTERVENTIONS:
Drug: Olinvacimab — Treatment with Olinvacimab and Pembrolizumab is to be continued until disease progression, the development of unacceptable toxicity or patient's withdrawal of consent. Maximum duration of treatment will be 35 cycles (approximately 2 years).
  Other Names: Pembrolizumab

SUMMARY:
The objective is to evaluate the efficacy and safety of Olinvacimab in combination with Pembrolizumab in patients with mTNBC.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients will complete informed consent form in written. During 2 weeks screening period, investigator will evaluate patient eligibility and if it meet with protocol, patient will enrolled. 1 cycle treatment is perform on D1, D8, D15 to inject Olinvacimab and Pembrolizumab, it can be repeated upto 35 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients ≥19 years old
2. Histologically proven mTNBC* irrespective of PD-L1 status.

   *Histological or cytological diagnosis of relapsed/metastatic TNBC. TNBC is defined by the negative expression of estrogen receptors (ER), progesterone receptors and human epidermal receptor-2 (HER2). If there is a pathology report of the metastasis, take the histopathology of the metastases as standard. Negative for ER and progesterone receptors is defined as the expression of ER and progesterone receptors in <1% of the tumor cells by immunohistochemistry (IHC). HER2-negative is defined as a score of 0 and 1+ by IHC, or IHC 2+ and fluorescence in situ hybridization (FISH) negative. If the HER2 test result is 0 or 1+ by IHC, FISH detection is optional, but the result must be negative.
3. Has provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.

   - Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut
4. Has measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
5. Has received at least one prior line of systemic therapy for metastatic or inoperable locally advanced TNBC. Patients who have failed adjuvant chemo within 12 months should be considered as fulfilling a line of systemic therapy.
6. No previous therapy with anti-VEGF, anti-VEGFR or anti-PD-1 antibody for their metastatic disease. The use of anti-VEGF, anti-VEGFR, anti-PD-1 or anti-PD-L1 antibody in neoadjuvant or adjuvant setting will be allowed if there was no progression of disease within 6 months after the completion of treatment.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
8. Adequate hematologic, renal, and hepatic function tests performed within 7 days prior to initiation of study treatment:

   * Hematologic tests

     * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
     * Platelets ≥ 100 x 109/L
     * Haemoglobin ≥ 9.0 g/dL (This must be met without packed red blood cell (pRBC) transfusion within the prior 2 weeks. Participants can be on stable dose of erythropoietin, e.g. ≥ approximately 3 months)
   * Blood coagulation tests

     * Prothrombin time (PT) ≤ 1.5 x Upper limit of normal (UNL)
     * Activated partial thromboplastin time (aPTT) ≤ 1.5 x UNL
   * Hepatic function tests

     * Total bilirubin ≤ 1.5 x UNL
     * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 x ULN (≤ 5 x ULN in case of liver metastasis)
   * Renal function test - Creatinine ≤1.5 × ULN or creatinine clearance (CrCl) ≥30 mL/min for patients with creatinine levels >1.5 × institutional ULN
9. HIV-infected participants must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease defined as:

   * Participants on ART must have a CD4+ T cell count >350 cells/mm3 at time of screening
   * Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 copies/mL or the lower limit of qualification (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks prior to screening
   * Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks prior to study entry (day 1)
10. Participants who are HBsAg positive are eligible if they have received HBV anti-viral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.

    * Note: Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.
    * Hepatitis B screening tests are not required unless:

      * Known history of HBV infection
      * As mandated by local health authority
11. Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.

    * Note: Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization.
    * Hepatitis C screening tests are not required unless:

      * Known history of HCV infection
      * As mandated by local health authority
12. The patient should provide written informed consent

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   - Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
2. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment
3. Treatment with systemic chemotherapy, hormonal therapy, immunotherapy or biologic therapy within 4 weeks or five half-lives (which is shorter) prior to the baseline visit
4. Has received prior radiotherapy within 2 weeks of start of study treatment. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 2-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease
5. Not recovered below National Cancer Institute (NCI) CTCAE (v5.0) Grade 1 or baseline from AEs due to previous therapy (patient with ≤ Grade 2 neuropathy or alopecia may be eligible)
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug
7. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. (Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ [e.g., breast carcinoma, cervical cancer in situ] controlled by curative therapy are not excluded).
9. Has a history of (non-infectious) pneumonitis/interstitial lung diseases that required steroids or current pneumonitis/interstitial lung disease
10. Has an active infection requiring systemic antibiotics
11. HIV-infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
12. Active psychiatric disorder (schizophrenia, major depressive disorder, bipolar disorder etc.) or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study. Treated depression with ongoing antidepressant medication is not an exclusion criterion
13. Female who is pregnant* or lactating and of childbearing potential who does not agree to a reliable and adequate method of contraceptiona.

    A women of childbearing potential (WOCBP) must agree to use contraception during the treatment period and for at least 6 months (for females) after the last dose of study treatment.

    aAdequate contraception allowed in this trial is as follows
    * Hormonal contraceptives such as combined oral contraceptive pill
    * Intrauterine devices (IUD) or the implantation of intrauterine system
    * Blockage methods (spermicides and condoms/spermicides and [vaginal] diaphragm for contraception, vaginal sponges or cervical cap)
    * Sterilization surgery such as tubal ligation in females *A WOCBP who has a positive urine pregnancy test (within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
14. Uncontrolled hypertension (systolic blood pressure [SBP]> 150 or diastolic blood pressure [DBP]> 90 mmHg) or seizure
15. Class III or IV heart failure by New York Heart Association (NYHA) classification
16. Requiring therapeutic anticoagulation treatment (prophylactic therapy with low-molecular weight heparin is allowed)
17. Serious Grade 4 venous thromboembolic event including pulmonary embolism
18. Moderate to severe proteinuria as demonstrated by urine dipstick for proteinuria ≥2+. For patients with ≥2+ proteinuria on dipstick urinalysis, a urine protein: creatinine (UPC) ratio will be determined, or a 24-hour urine collection will be done. Patients with a UPC ratio <1 or a 24-hour urine protein <1 gram are eligible.
19. History of abdominal fistula or gastrointestinal perforation, or serious GI bleeding within 6 months
20. History of severe arterial thromboembolic event within 12 months of start of study drug
21. Major surgery within 4 weeks prior to initiation of study treatment. (If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention).
22. A known history of severe hypersensitivity (≥Grade 3) to study drugs and/or any of its excipients.
23. Has had an allogenic tissue/solid organ transplant.
24. Unable to participate in the trial according to the investigator's decision.
25. Have received a live vaccine within 30 days prior to enrollment. Seasonal flu vaccines that do not contain live virus are permitted
26. Have had a serious or non-healing wound, ulcer, or bone fracture within 28 days prior to enrollment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Baseline upto 24 months
  ORR is defined as the proportion of subjects who achieve a best overall response (BOR) of complete response (CR) or partial response (PR). RECIST 1.1 will be used to determine ORR and patients with no post baseline tumor assessments, will be classified as non-responders

SECONDARY OUTCOMES:
Duration of response (DOR) | Baseline upto 24 months
  DOR is defined as the time between the date of first response (CR or PR) according to RECIST 1.1 to the date of first disease progression, or death due to any cause, whichever occurs first.
Disease control rate (DCR) | Baseline upto 24 months
  DCR is defined as the proportion of subjects who achieve CR, PR, or stable disease (SD) according to RECIST 1.1.
Progression-free survival (PFS) | Baseline upto 24 months
  PFS time is defined as the time from the start date of the study drug administration to date of the first disease progression according to RECIST 1.1, or death due to any cause, whichever occurs first.
Overall survival (OS) | Baseline upto 24 months
  OS time is defined as the time from the start date of the study drug administration to the date of death due to any cause.

OTHER OUTCOMES:
ORR evaluated by iRECIST criteria: | Baseline upto 24 months
  ORR will be evaluated based on iRECIST criteria in the FAS.
DOR evaluated by iRECIST criteria: | Baseline upto 24 months
  DOR will be evaluated based on iRECIST criteria in the FAS.
DCR evaluated by iRECIST criteria: | Baseline upto 24 months
  DCR will be evaluated based on iRECIST criteria in the FAS.
PFS evaluated by iRECIST criteria: | Baseline upto 24 months
  PFS will be evaluated based on iRECIST criteria in the FAS.
OS evaluated by iRECIST criteria: | Baseline upto 24 months
  OS will be evaluated based on iRECIST criteria in the FAS.
Pharmacodynamic evaluation | Baseline upto 24 months
  Change in concentration of serum biomarkers
Exome sequencing of tumor tissue | Screening visit
  The descriptive information of tumor tissue with mutation
Immune suppression by level of circulating MDSC population | Baseline upto 24 months
  The percent change of MDSC compared to baseline (before treatment on day 1 of cycle 1) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Beecroft, Ph.D, MD, Principal Investigator — Hollywood Private Hospital, Australia; Dhanusha Sabanathan, Ph.D, MD, Principal Investigator — Macquarie University, Australia; Brenton Seidl, Ph.D, MD, Principal Investigator — University of Sunshine Coast, Australia; Daphne Day, Ph.D, MD, Principal Investigator — Monash Medical Centre, Australia
Locations (1):
- Hollywood Private Hospital, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No